CLINICAL TRIAL: NCT05367843
Title: A Phase 1, Dose Ranging Study Assessing the Safety, Tolerability, Immunogenicity of Vaccine Candidate PRIME-2-CoV_Beta, Orf Virus Expressing SARS-CoV-2 Spike and Nucleocapsid Proteins (ORFEUS Study)
Brief Title: A Study Assessing the Safety, Tolerability, Immunogenicity of COVID-19 Vaccine Candidate PRIME-2-CoV_Beta, Orf Virus Expressing SARS-CoV_2 Spike and Nucleocapsid Proteins
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Speransa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: D1701-VrV-101; 2021-005219-30 (EudraCT Number)
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Coronavirus; COVID-19; PRIME-2-CoV_Beta
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — PRIME-2-CoV_Beta COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A-Cohorts: Pre-vaccinated (Experimental): Participants aged 18-55 years who have been pre-vaccinated against COVID-19 with at least two doses of a SARS-CoV-2 mRNA vaccine will be assigned to five groups that receive increasing doses of PRIME-2-CoV_Beta (two doses, 28 days apart).
  Interventions: Drug: PRIME-2-CoV_Beta
- A-Cohorts: SARS-CoV-2 Vaccine-naïve (Experimental): Participants aged 18-55 years who are SARS-CoV-2 vaccine-naïve will receive one preferred dose level of PRIME-2-CoV_Beta that has been identified as optimal in pre-vaccinated A-Cohorts (two doses, 28 days apart).
  Interventions: Drug: PRIME-2-CoV_Beta
- B-Cohorts: Pre-vaccinated elderly (Experimental): Elderly participants aged 65-85 years who have been previously vaccinated against COVID-19 with at least two doses of a SARS-CoV-2 mRNA vaccine will be assigned to three groups to receive previously identified doses of PRIME-2-CoV_Beta (two doses, 28 days apart).
  Interventions: Drug: PRIME-2-CoV_Beta

INTERVENTIONS:
Drug: PRIME-2-CoV_Beta — Intramuscular (IM) injection

SUMMARY:
PRIME-2-CoV_Beta is the first clinical candidate based on the attenuated 2nd generation Orf virus (ORFV) vaccine platform which encodes for the structural spike (S)- and nucleocapsid (N) protein of SARS-CoV-2. The aim of the multivalent vaccine is to broaden the specific immune response against SARS-CoV-2 and to increase the probability of cross-protection against emerging variants.

DETAILED DESCRIPTION:
The Phase 1 dose-finding study (ORFEUS) will assess the safety, tolerability and immunogenicity of a two-dose regimen (28-days apart) of PRIME-2-CoV_Beta administered by intramuscular (IM) route in adult participants.

In the first part, the safety and immunogenicity of increasing doses of PRIME-2-CoV_Beta will be assessed in adult healthy participants aged 18 to 55 years who have been vaccinated against COVID-19 with at least two doses of a SARS-CoV-2 mRNA vaccine (i.e. primary sequence with or without booster vaccination, subsequently referred to as "pre-vaccinated"). In addition, one dose level which has been identified as optimal will be assessed in a small cohort (12 participants) of participants 18 to 55 years of age who are SARS-CoV-2 vaccine-naïve.

In addition, three dose levels identified in pre-vaccinated participants will be further evaluated for safety and immunogenicity in pre-vaccinated elderly participants aged 65-85 years (B-cohorts).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between the ages of 18 and 55 years, (A-cohorts), and 65 and 85 years (B-cohorts), inclusive at study entry.
2. Body mass index (BMI) over 19 kg/m^2 and under 32 kg/m^2 and weight at least 50 kg at study entry.
3. Healthy participants who are determined by medical history, physical examination, and clinical judgment of the Investigator to be eligible for inclusion in the study.

   Note: Healthy participants may have stable pre-existing disease defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment.
4. Able to give personal signed informed consent and willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, and other study procedures.
5. Participants must agree not to be vaccinated with any SARS-CoV-2 vaccine, starting after Visit 0 and continuously until 6 months after receiving the first study immunization.
6. Participants who have previously received at least two vaccinations with a licensed SARS-CoV-2 mRNA vaccine (Spikevax/Moderna and/or Comirnaty/Pfizer administered as two-dose primary series with or without booster vaccination[s]) with the last vaccination having occurred at least 3 months prior.
7. Participants who are SARS-CoV-2 vaccine-naïve (applies to vaccine-naïve group of Cohort A only):

   1. Currently not working in occupations with high risk of exposure to SARS-CoV-2 (e.g., healthcare worker, emergency response personnel) (vaccine-naïve group of Cohort A only).
   2. No previous vaccination with any SARS-CoV-2 vaccine (vaccine-naïve group of Cohort A only).
8. If the participant is a woman of child bearing potential (WOCBP) must:

   1. have a negative beta-human chorionic gonadotropin (hCG)-urine test at Visit 0 and Visit 1.
   2. agree to practice a highly effective form of contraception for at least 14 days prior to study vaccination and continuously until a minimum of 28 days after receiving the last immunization.
   3. agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study, starting after Visit 0 and continuously until 28 days after receiving the last immunization.

   Note: Women that are postmenopausal or permanently sterilized will be considered as not having reproductive potential.
9. Men who are sexually active with a WOCBP and have not had a vasectomy must agree to practice a highly effective form of contraception with their female partner during the study, starting from Visit 1 (pre-dose) and continuously until a minimum of 28 days after receiving the last immunization.
10. Men must be willing to refrain from sperm donation, starting from Visit 1 (pre-dose) and continuously until a minimum of 28 days after receiving the last immunization.

Exclusion Criteria:

1. SARS-CoV-2 nucleic acid amplification test (NAAT)-positive pharyngeal swab within 24 hours before receipt of study vaccine.
2. Previously NAAT-confirmed COVID-19 within the last 2 months prior to vaccination.
3. Participants who are taking medications which may prevent or treat COVID-19.
4. Participants who received convalescent serum or prior therapeutic antibodies against SARS-CoV-2 in a period of 6 months.
5. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study vaccine(s).
6. Current clinical or microbiological diagnosis of COVID-19, including active respiratory or non-respiratory symptoms associated with COVID-19 disease (i.e. symptomatic COVID-19 disease).
7. Any respiratory illness deemed clinically relevant by the investigator within the past month OR hospitalization >24 hours for any reason within the past month.
8. History of or current cardiac disease, including but not limited to individuals with uncontrolled hypertension (defined as grade 1 hypertension or higher as per ISH guidelines with or without antihypertensive medication), congenital structural heart diseases, myocarditis and/or pericarditis, coronary heart disease (with/without angina pectoris) or myocardial infarction.
9. Individuals with myocarditis after mRNA vaccination, or individuals with AEs after mRNA-vaccination that are in nature and severity beyond the common AEs that can be expected.
10. Individuals at high risk for severe COVID-19, including those with any of the following risk factors: cancer; chronic kidney disease; chronic obstructive pulmonary disease (COPD); immunocompromised state (weakened immune system) from solid organ transplant; rheumatologic or autoinflammatory conditions requiring immunosuppressive medication, malignancies; obesity (BMI of 32 or higher); serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies; sickle cell disease; insulin-dependent type 2 diabetes mellitus.
11. Anticipating the need for immunosuppressive treatment within the next 6 months.
12. Any screening hematology and/or blood chemistry laboratory value outside normal range (defined as ≥Grade 1 abnormality) and deemed clinically relevant by the investigator.

    Note: Except bilirubin, participants with any stable Grade 1 abnormalities may be considered eligible at the discretion of the Investigator.
13. Chronic immunosuppressive therapy (defined as ≥14 days), including cytotoxic agents, systemic corticosteroids exceeding 10mg/d prednisone equivalent, disease-modifying antirheumatic drugs [DMARDs]) or any other immunomodulating agents within the last 3 months or planned receipt throughout the study.

    Note: If systemic corticosteroids have been administered short-term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
14. Receipt of blood/plasma products or immunoglobulin from 60 days before study vaccine administration or planned receipt throughout the study.
15. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
16. Individuals with a history of or active autoimmune disease requiring therapeutic intervention.

    Note: subjects with vitiligo or thyroid disease on stable dose thyroid hormone replacement may be enrolled at the discretion of the investigator.
17. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
18. History of human immunodeficiency virus (HIV), known seropositivity or active infection with HIV.
19. History of known seropositivity for or evidence of active viral infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).

    Exception: Participants who are seropositive because of HBV vaccine are eligible. Participants who had HCV but have received an antiviral treatment and show no detectable HCV viral deoxyribonucleic acid (DNA) for 6 months are eligible.
20. Known history of active or latent tuberculosis (bacillus tuberculosis).
21. Any concomitant serious health condition or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior, which, in the opinion of the Investigator, would place the participant at undue risk from the study.
22. Has received a live vaccine within 28 days of planned start of study vaccinations (i.e. 28 days before the first and after the last vaccination).
23. If a participant has contraindication to IM injections according to investigator's assessment or received therapeutic-intensity anticoagulation for a thromboembolic event within a period of 60 days before vaccination.

    Note: stable long-term prophylactic-dose anticoagulation is allowed.
24. Participants with prolonged exposure to sheep or goats (e.g., shepherds, sheep farmer).
25. Pregnant and/or nursing women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with solicited local reactions at the injection site | Up to 7 days after first immunization (Day 1 up to 8)
  Solicited local reactions are described as pain, erythema/redness and induration/swelling.
Number of participants with solicited local reactions at the injection site | Up to 7 days after second immunization (Day 29 up to 36)
  Solicited local reactions are described as pain, erythema/redness and induration/swelling.
Number of participants with solicited systemic reactions | Up to 7 days after first immunization (Day 1 up to 8)
  Solicited systemic reactions are described as nausea, vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and fever.
Number of participants with solicited systemic reactions | Up to 7 days after second immunization (Day 29 up to 36)
  Solicited systemic reactions are described as nausea, vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and fever.
Number of participants who experience at least one unsolicited Treatment-emergent Adverse Event (TEAE) | Day 1 up to Day 57

SECONDARY OUTCOMES:
Geometric mean of SARS-CoV-2-specific serum neutralizing titers against ancestral and variant SARS-CoV-2 strains at each time point | Up to 6 months
Geometric Mean-fold Rise (GMFR) of SARS-CoV-2-specific serum neutralizing titers against ancestral and variant SARS-CoV-2 strains from baseline to each subsequent timepoint | Up to 6 months
Number of participants who achieve ≥ 4-fold rise from baseline in SARS-CoV-2-specific serum neutralizing titers against ancestral and variant SARS-CoV-2 strains from baseline to each subsequent timepoint | Up to 6 months
Geometric Mean Concentration (GMC) of SARS-CoV-2-spike and nucleocapsid-protein specific binding antibody levels from baseline to each subsequent time point | Up to 6 months
Geometric Mean-fold Rise (GMFR) of SARS-CoV-2-spike and nucleocapsid-protein specific binding antibody levels from baseline to each subsequent time point | Up to 6 months
Number of participants who achieve ≥ 4-fold rise in SARS-CoV-2-spike and nucleocapsid-protein specific binding antibody levels from baseline to each subsequent time point | Up to 6 months
Recommended Phase 2 Dose (RP2D) of PRIME-2-CoV_Beta | Up to 12 months
  RP2D based on an integrated analysis of overall safety and immunogenicity endpoints (change in SARS-CoV-2-specific serum neutralizing titers and SARS-CoV-2-spike protein-specific and -nucleocapsid protein-specific binding antibody levels.
Safety and tolerability assessed as incidence of changes from baseline in clinical laboratory values, vital Signs, and Electrocardiograms (ECGs) | Up to 6 months
  Endpoint is assessed as a composite of clinical lab values, vital signs, and ECGs.
Number of participants with solicited local reactions at the injection site | Up to Day 15
  Solicited local reactions are described as pain, erythema/redness and induration/swelling.
Number of participants with solicited systemic reactions | Up to Day 15
  Solicited systemic reactions are described as nausea, vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and fever.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Accel Research Sites (ARS) - DeLand Clinical Research Unit, Florida City, Florida
  - Cedar Crosse Research Center, Chicago, Illinois
  - AMR - Center for Pharmaceutical Research - Kansas City, Kansas City, Missouri
  - Caroline Institute for Clinical Research, Fayetteville, North Carolina
  - Cedar Health Research - DFW-East, Dallas, Texas
- Germany (2):
  - Clinical Research Center Hannover, Hanover
  - Ludwig-Maximilians-University Munich (LMU), Munich

REFERENCES:
- [Derived] Klinkardt U, Schunk M, Ervin J, Schindler C, Sugimoto D, Rankin B, Amann R, Monti M, Kutschenko A, Schumacher C, Huber K, Zeder A, Heikkila N, Didierlaurent AM, Schwarz SE, Derouazi M. A novel orf virus vector-based COVID-19 booster vaccine shows cross-neutralizing activity in the absence of anti-vector neutralizing immunity. Hum Vaccin Immunother. 2024 Dec 31;20(1):2410574. doi: 10.1080/21645515.2024.2410574. Epub 2024 Oct 14. PMID 39397784